CLINICAL TRIAL: NCT05034172
Title: Biomarker Research in Inherited Movement Disorders
Acronym: BIOMOV
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210069
Record Dates: First submitted 2021-06-17; First posted 2021-09-05 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Inherited Movement Disorders; Spinocerebellar Ataxias; Hyperkinetic Disorders
MeSH Terms: conditions — Spinocerebellar Ataxias; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples (optional) : blood sample, skin biopsy, excreta collection (saliva, urine, feces), cerebrospinal fluid collection (if Lumbar Puncture in standard care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical follow-up — Clinical Follow-up:
  demographic data and history,
  * Retrospective interview (collection of data useful for genetic studies): -disease history (for patients only);
  * Family history - Neurological examination:
  * Diagnosis Clinical examination;
  * Rating scales specific to the pathology under investigation;
  * Cerebral MRI (optional)
  * Biological samples (optional)

SUMMARY:
Inherited movement disorders are rare conditions, whose cumulative prevalence are in the order of 5-10/100,000 inhabitants, in most cases progressive and can lead to a significant loss of autonomy after one or more decades of evolution. They include spinocerebellar ataxias and hyperkinetic disorders (dystonias, choreas, tremor, parkinsonism and myoclonus with variable combination of those, or more complex alteration of movements). The existence of the National Reference Centre (CMR) for Rare Diseases (CMR Neurogenetics, devoted to ataxias and spastic paraparesis, dystonia and rare movement disorders and CMR Huntington, devoted to Huntington Disease) has allowed a more integrated vision of these diseases. This is illustrated, in the same family, by the occurrence of different clinical expressions of spinocerebellar ataxias and hyperkinetic disorders that share the same genetic background. Conversely, different causal mutations within the same gene may have very different ages at onset and a wide range of clinical expression, and the spectrum of new phenotypes linked to a single gene is still expanding . Many ataxia and dystonia genes are involved in similar pathways. There are numerous arguments supporting a share pathogenesis including synaptic transmission and neurodevelopment .

BIOMOV project aims to :

1. establish the clinical spectrum and natural history of these diseases,
2. understand the role of genetic and familial factors on the phenotype,
3. elucidate the molecular basis of these disorders and evaluate diagnostic strategies involving molecular tools for clinical and genetic management,
4. develop multimodal biomarkers both for physiopathological studies and for accurate measures of disease progression,
5. develop trial ready cohorts of well characterized genetic patients,
6. test new therapies either symptomatic or based on pathophysiological mechanisms.

DETAILED DESCRIPTION:
Inherited movement disorders are rare conditions, whose cumulative prevalence are in the order of 5-10/100,000 inhabitants, in most cases progressive and can lead to a significant loss of autonomy after one or more decades of evolution. They include spinocerebellar ataxias and hyperkinetic disorders (dystonias, choreas, tremor, parkinsonism and myoclonus with variable combination of those, or more complex alteration of movements). The existence of the National Reference Centre (CMR) for Rare Diseases (CMR Neurogenetics, devoted to ataxias and spastic paraparesis, dystonia and rare movement disorders and CMR Huntington, devoted to Huntington Disease) has allowed a more integrated vision of these diseases. This is illustrated, in the same family, by the occurrence of different clinical expressions of spinocerebellar ataxias and hyperkinetic disorders that share the same genetic background. Conversely, different causal mutations within the same gene may have very different ages at onset and a wide range of clinical expression, and the spectrum of new phenotypes linked to a single gene is still expanding .

any ataxia and dystonia genes are involved in similar pathways. There are numerous arguments supporting a share pathogenesis including synaptic transmission and neurodevelopment .

Overall, there are a number of arguments for a shared genetic approach and biomarkers research for these inherited movement disorders:

* Evidence from a clinico-genetic approach: A combination of several movement disorders is often observed in the same patient with causative mutation in either genetic groups of spinocerebellar degenerations, dystonias or choreas.
* Evidence from neuroimaging: the current concept of networks disorders underlies the pathophysiology of these hyperkinetic movement disorders. Variable combination of functional and/ or structural alterations of the cerebello-thalamo-cortical, cortex-basal ganglia and corticospinal networks, and their complex interactions have been described in ataxias ,dystonia choreas and more complex disorders.
* Genetic diagnosis: deciphering diagnosis with wide range of phenotypes Even in times of next generation sequencing covering exomes and genomes, diagnosing spinocerebellar degenerations, dystonia and other hyperkinetic disorders remains a challenge as: i) the causative gene remains to be identified for a substantial share those disorders; the pathogenicity of variants of unknown significance in known and potential novel disease genes often requires time-consuming functional analyses not available on a routine basis; ii) in many countries, including France, access to diagnostic whole exome and whole genome sequencing is still limited; iii) the proportions of abnormal expansions not seen in exome studies are frequent in spinocerebellar degenerations and need a technological development to identify them. Analysis of familial forms revealed a great heterogeneity of the phenotype within the same family in terms of age at onset, severity and clinical presentation. Moreover, this phenotypic variability is not explained only by the genetic heterogeneity but also by the underlying frequent exonic or intronic expansions of triplet or more complex repeats, and more recently by the discovery of genetic modifiers ; iv) for dystonia and hyperkinetic disorders, some of those disorders also include nonmovement disorders neurological (e.g. intellectual deficiencies, hypotonia at birth, immature motor control, deafness, visual defects) and non-neurological (dysmorphological features) symptoms and the movement disorders panels do not always include the genes involved in developmental disorders; v) among the dominantly inherited forms such as Huntington disease, the access to genetic testing procedures allows early preventive therapeutic interventions in premanifest individuals. There is a lack of clinical evaluation to tackle the efficiency of treatment and the need for biomarker development.
* Natural history and prognosis: need for quantitative, reproducible markers, sensitive to evolution Biomarkers search is ongoing in those pathologies. They are valuable in assisting diagnosis, have prognostic value, quantify disease progression and serve as outcome parameters in clinical trials.

These elements demonstrate the need to develop quantitative tools that are easy to use, reproducible and sensitive to disease progression in order to accurately determine the natural history of the disease. This lack of systematic knowledge impedes diagnosis, patient counselling and therapy development.

Overall: Identification of the underlying gene and its pathogenic changes or variant(s) contributes to precise diagnosis, genetic counselling and follow-up. Advances in molecular genetics have highlighted the genotypic complexity, justifying the need for rigorous clinical and para-clinical evaluation to establish relevant phenotype-genotype correlations. In dystonia and in spinocerebellar degenerations attempts have been made to classify the genes involved.

Molecular genetic analysis will make it possible to specify the correlations between phenotype and genotype in order to propose rational molecular diagnostic strategies based on the frequency and nature of mutations, taking into account the phenotype. Genetic analyses will have an impact in terms of public health since they will serve as a basis for guiding requests for molecular analyses in these pathologies. In addition, recent advances in therapeutic trials will need the careful selection of participants, mostly based on biomarkers, for successful testing of new therapeutical agents. Therefore, it seems essential that this cohort of patients be supplemented by a collection of biological material for genetic research.

BIOMOV project aims to : 1) establish the clinical spectrum and natural history of these diseases, 2) understand the role of genetic and familial factors on the phenotype, 3) elucidate the molecular basis of these disorders and evaluate diagnostic strategies involving molecular tools for clinical and genetic management, 4) develop multimodal biomarkers both for physiopathological studies and for accurate measures of disease progression, 5) develop trial ready cohorts of well characterized genetic patients, 6) test new therapies either symptomatic or based on pathophysiological mechanisms.

It is crucial to be able to establish a large cohort of patients whose genotype will be specified. Follow-up of patients at different stages of the disease will make it possible to collect the natural history of the disease in a descriptive manner, with prospects for patient management, since the prognosis in terms of loss of autonomy or disability will be better specified. However, the main interest of the proposed clinical follow-up is to be able to quantitatively describe the progression of the main neurological diseases. These data are absolutely essential for the future implementation of therapeutic trials. The number of patients likely to be recruited and followed up a unique resource for such a project

ELIGIBILITY:
Inclusion Criteria:

Common inclusion criteria for all participants:

- - Affiliated with a social security system or beneficiary of such a regime

Group of patients:

Any patient with inherited hyperkinetic movement disorders can be included in the study according to the following criteria:

Woman or man;

* Clinical diagnosis of inherited hyperkinetic movement disorders with or without a genetic diagnosis
* With or without familial history of the disease
* Age ≥ 7 years;
* Signed Informed consent by the patient or both of holders of the parental authority for minors, or by the le;gal guardian for adults under guardianship

Group of at-risk individuals:

* Woman or man;
* Age ≥ 18 years old;
* A first-degree relative of a patient with inherited hyperkinetic movement disorders
* OR a carrier of an identified pathogenic variant or expansion in one of the pathological gene variant involved in one of these diseases;
* Normal neurological examination; according to disease specific scales
* Signed Informed consent by the subject or by the legal guardian for adults under guardianship

Group of healthy controls:

* Woman or man;
* Aged ≥ 18 years old;
* Free of known neurological pathology;
* No significant neurological symptoms;
* Signed Informed consent by the subject

Common inclusion criteria for elective participant for skin biopsy (optional): - Age ≥10 ans

* Ability to undergo a skin biopsy

Common inclusion criteria for elective participant for MRI examination (optional): - Ability to undergo a MRI.

Exclusion Criteria:

Absolute criteria for non-inclusion for all groups:

- Person deprived of their liberty by judicial decision

Contra-indications to MRI examination* (optional): metallic implant, pacemaker, artificial heart valve, brain vascular malformation, aneurysm clips, exposed by metallic fragments, artificial implants, peripheral or neuronal stimulator, insulin pump, intravenous catheter, epilepsy, metallic contraceptive device, claustrophobia,

Contra-indication to skin biopsy (optional):

* Taking anticoagulant or antiplatelet medication (see above),
* History of hemostasis disorders,
* Presence of hemorrhagic risk verified by a coagulation test

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with hyperkinetic movement disorders
  * At risk individuals (gene mutation carriers) with inherited hyperkinetic movement disorders
  * Healthy controls to allow variant classification and establish normal values for scales
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2031-08-25 (Estimated); Study Completion 2031-08-25 (Estimated)

PRIMARY OUTCOMES:
Genetic entities among rare movement disorders: Pathology characterization (clinical spectrum) and its natural history: clinical Biomarkers | 10 years
  Comparison of clinical biomarkers at different disease stages compared to controls.
Genetic entities among rare movement disorders: Pathology characterization (clinical spectrum) and its natural history : genetic Biomarkers | 10 years
  Comparison of genetic biomarkers at different disease stages compared to controls.
Genetic entities among rare movement disorders: Pathology characterization (clinical spectrum) and its natural history : biological and/or imaging Biomarkers | 10 years
  Comparison of biological and/or imaging biomarkers at different disease stages compared to controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpetrière, Paris, France